CLINICAL TRIAL: NCT04852627
Title: Effect of Brisk Walking on Primary Dysmenorrhea Among Medical Students
Brief Title: Effect of Brisk Walking on Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M D 59/2021
Record Dates: First submitted 2021-04-17; First posted 2021-04-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Dysmenorrhea Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): Will brisk walk 30 minutes 3 times weekly
  Interventions: Behavioral: Brisk walking
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Brisk walking — Walking
  Arms: Exercise group

SUMMARY:
Dysmenorrhea is a common problem in women. Exercise is commonly cited as a possible remedy. We will measure the effect of brisk walking on primary dysmenorrhea among medical students.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18-25
* regular menstrual cycles

Exclusion Criteria:

* Marriage or previous sexual activity
* medical disorders
* previous abdominal or pelvic surgery
* skeletal disorders
* hormonal or psychiatric treatment
* atheletes

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Must be female
Enrollment: 170 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Dysmenorrhea score | 3 months
  WaLIDD (working ability, location, intensity, days of pin, dysmenorrhea)score for dysmenorrhea. Least is 0, highest is 12. The higher the score, the worse dysmenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Maii Nawara, MD, Principal Investigator — Ain Shams University
Locations (1):
- AinShams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available with the principal investigator and will be shared if requested